19-10-2018

(S1)

## Informed consent for participation in a health science research project.

Research project title: MELADERM-trial: Melatonin cream against acute radiation dermatitis in patients with early breast cancer: a pivotal phase 2, double-blind, randomized, placebo-controlled trial

## **Declaration by the subject:**

EudraCT nr.: 2018-001705-91

I have received written and oral information and I know enough about the purpose, method, advantages and disadvantages to say yes to participate.

I know it's voluntary to participate and that I can always withdraw my consent without losing my current or future rights to treatment.

I agree to participate in the research project and have received a copy of this consent sheet as well as a copy of the written information about the project for its own use.

| Subject name: | |
|---|---|
| Date: Signature: | |
| Do you want to be informed about the results of the research pro | oject and any consequences for you?: |
| Yes (mark with x) No (mark with x) | |
| Declaration of the person providing information: | |
| I declare that the subject has received oral and written informati | on about the trial. |
| In my conviction, sufficient information has been provided for a control of the person who provided information: | decision to participate in the trial. |
| Date: Signature: | |

Project identification: EudraCT nr.: 2018-001705-91